CLINICAL TRIAL: NCT03514836
Title: A Phase I/II, Clinical Trial to Evaluate the Safety and Immune Activation of the Combination of DCVAC/PCa, and ONCOS-102, in Men With Advanced Metastatic Castration-resistant Prostate Cancer.
Brief Title: A Phase I/II, Safety Clinical Trial of DCVAC/PCa and ONCOS-102 in Men With Metastatic Castration-resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: insufficient accrual
Sponsor: SOTIO a.s. (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP015
Record Dates: First submitted 2018-04-11; First posted 2018-05-02 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Castration-resistant Prostate Cancer
Keywords: Castrate-resistant
MeSH Terms: interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Open label combination treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DCVac and ONCOS-102 (Experimental): ONCOS-102 is given intra-tumor up to 4 times, cyclophosphamide is given prior to the first dose of ONCOS-102 and at the fifth week of treatment DCVac is given sc every 21-28 days for up to 10 doses
  Interventions: Biological: DCVac/PCa; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: DCVac/PCa — Oncolytic adenovirus containing immunostimulatory cytokine granulocyte-monocyte colony-stimulating factor (GM-CSF). This is an experimental therapy.
  DCVac/Pca consists of activated autologous dendritic cells. This is an experimental therapy.
  Other Names: ONCOS-102
Drug: Cyclophosphamide — immunomodulatory medication given around the ONCOS-102 dosing

SUMMARY:
This clinical trial is to evaluate the safety of the combination of DCVAC/PCa with ONCOS-102 in men with castration-resistant advanced metastatic prostate cancer, who have progressed following initial therapy with either hormones (e.g. abiraterone and enzalutamide) or chemotherapy.

Male patients with castration-resistant advanced metastatic prostate cancer, who have progressed following initial therapy with either All patients must have at least one readily accessible soft tissue/nodal tumor lesion (for intra-tumoral application of ONCOS-102 and biopsy.

DETAILED DESCRIPTION:
Study Description:

* All patients who fulfill all eligibility criteria will undergo a leukapheresis procedure.
* ONCOS-102 administration will start within 3 weeks of leukapheresis at Week 5 (35 days since baseline +/- 2 days), and 3 further doses will be administered on a weekly basis
* Cyclophosphamide A priming bolus dose of CPO (300 mg/m2 intravenously) will be given 1-3 days before the first (Week 5) and the fifth (Week 14) of ONCOS-102 administration.
* DCVAC/PCa therapy will start 6 weeks after leukapheresis at Week 8. DCVAC/PCa will be administered subcutaneously in cycles, always on Day 1 (+/- 3 days) of the corresponding cycle.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Radiographically documented metastatic disease with evidence of disease progression Laboratory parameters per protocol
* Surgically or medically castrate
* Patients who have progressed following:
* a. at least initial therapy (chemotherapy or treatment with a hormonal agent known to impact survival such as abiraterone and enzalutamide); or
* b. one first-line chemotherapy regimen and one additional hormonal agent known to impact survival such as abiraterone and enzalutamide; or
* c. failure of two lines of chemotherapy; or
* d. failure of pre-chemotherapy abiraterone or enzalutamide and subsequent chemotherapy

Exclusion Criteria:

* Patients with neuroendocrine or small cell cancer of the prostate 2. History of other malignant disease (with the exception of the primary prostate cancer and non-melanoma skin tumors) in the past 5 years Pre-defined co-morbidities
* Administration of experimental therapy within the last 4 weeks before start of screening
* Treatment with immunotherapy within the last 3 months before start of screening
* Treatment with radiopharmaceutical drugs within 8 weeks before start of screening
* Receipt of oncolytic virus treatment or vaccination with a live virus within 4 weeks of study start
* History of organ transplantation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate Cancer
Enrollment: 5 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 96 months
  PFS measured by modifications to the RECIST 1.1. PFS is defined as the time from the first dose of SoC therapy administered to tumor progression or death from any cause.

SECONDARY OUTCOMES:
Overall Survival | 96 months
  Defined as the time from Baseline visit to the date of death for any cause
Safety | 96 months
  Reports of adverse events, serious adverse events, lab abnormalities utilizing NCI CTCAE v.4.033
Time to Progression-PSA | 96 months
  demonstrated by rising PSA as defined by the Prostate Cancer Workging Group2
Radiographic Progression- free survival | 96 months
  composite assessment of progression of bone lesions, soft-tissue lesions or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Roman Korolkiewicz, MD, PhD, Study Director — Sotio as
Locations (1):
- Fakultní nemocnice v Motole, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided